CLINICAL TRIAL: NCT01585831
Title: Psychological and Motor Effects of Testosterone Therapy in Adolescents With XXY/Klinefelter Syndrome
Brief Title: Study of Psychological and Motor Effects of Testosterone in Adolescents With XXY/Klinefelter Syndrome
Acronym: TestoXXY/KS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); Children's Hospital Colorado (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0874; 1K23NS070337 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-26 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Klinefelter Syndrome; XXY Syndrome
Keywords: Klinefelter syndrome; XXY syndrome; Sex Chromosome Abnormality; Testosterone replacement therapy
MeSH Terms: conditions — Klinefelter Syndrome; Sex Chromosome Aberrations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone gel 1% (Experimental): Testosterone gel 1% applied to skin once per day for 1 year. Starting dose 1.25mL per day, titrated in 1.25mL increments for 1st 6 months of study after each study visit up to maximum of 5.0mL per day. Titration based on testosterone levels with target level in mid-range of normal for Tanner stage.
  Interventions: Drug: Testosterone gel 1%
- Placebo gel (Placebo Comparator): Placebo gel applied to skin once per day for 1 year. Starting dose 1.25mL per day. Dose randomly adjusted in 1.25mL increments for 1st 6 months of study after each study visit up to maximum of 5.0mL per day.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Testosterone gel 1% — Testosterone gel will be administered on a daily basis. The gel will be dispensed in a syringe, and the specific amount of gel to be applied each day will be determined by the study endocrinologist after reviewing labs.
  Other Names: Androgel 1%
  Arms: Testosterone gel 1%
Drug: Placebo gel — The placebo gel will be administered on a daily basis. The gel will be dispensed in a syringe, and the specific amount of gel to be applied each day will be determined by the study endocrinologist.
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to determine if testosterone replacement therapy leads to changes in psychological factors and/or motor skills in adolescent males with 47,XXY (also called Klinefelter syndrome). This study will also evaluate whether certain genetic factors of the X chromosome affect the psychological or motor features of XXY/Klinefelter syndrome.

DETAILED DESCRIPTION:
Klinefelter syndrome (47,XXY) is the most common chromosomal abnormality in humans and occurs in approximately 1 in 650 males. Testosterone deficiency develops during adolescence in the majority of individuals with XXY. However, there are no previous studies that evaluate the psychological and motor effects of testosterone replacement therapy in adolescents with XXY.

The study researchers are interested in learning if testosterone therapy initiated in early puberty in XXY (KS) will lead to improvements in psychological and/or motor skills. They are also interested in learning if genetic variations of the androgen receptor gene or the parent-of-origin of the extra X chromosome influence the response to testosterone therapy.

Specific psychological factors to be studied include verbal and nonverbal cognitive skills, attention, executive function (organization, problem-solving skills, inhibition), anxiety, language, self-esteem, and other behavioral factors. Motor skills to be studied include gross and fine motor skills, motor coordination, and motor planning.

Participants in the study will be randomized to one of two treatment groups, receiving either testosterone gel or placebo, for 12 months. 60% of the study group will receive testosterone, and 40% will receive placebo.

The research participants, parents/caregivers, and the members of the study team will be blinded to the treatment group, and will not know whether they are receiving testosterone gel or placebo treatments.

The supervising endocrinologist for the study will not be blinded and will know which patients are in the testosterone and placebo groups. This will allow him to monitor results to determine if participants in the placebo group may develop a significant need for testosterone therapy during the study period. If this occurs, the patient will be switched to the testosterone group and will continue to be monitored in the study.

All participants will be evaluated at the beginning of the study and at 1, 3, 6, and 12 months. Travel costs are included. Evaluations will include a combination of psychological and motor skills testing, questionnaires completed by the parent/caregiver and study participant, physical examinations, and blood draws for safety monitoring and genetic studies.

Participation in the trial will last one year and includes 5 clinic visits to the eXtraordinarY Kids Clinic at Children's Hospital Colorado in Denver.

ELIGIBILITY:
Inclusion Criteria:

* Males with 47,XXY
* Participants must be in early puberty (Tanner stage II-III)
* Age 8 - 18 will be considered, but eligibility will be determined by review of laboratory results, bone age X-ray, and physical examination to determine stage of puberty
* All racial and ethnic groups

Exclusion Criteria:

* Other genetic variations of Klinefelter syndrome (48,XXXY, 48,XXYY, 49,XXXXY). The investigator has other studies for these groups and we encourage interested individuals with these disorders to contact us about other available studies.
* 47,XXY plus another genetic disorder
* Non-English speaking individuals (because the psychological tests are administered in English)
* Participants with a medical history of blood clotting problems, blindness, deafness, or cancer

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Tartaglia, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Davis SM, DeKlotz S, Nadeau KJ, Kelsey MM, Zeitler PS, Tartaglia NR. High prevalence of cardiometabolic risk features in adolescents with 47,XXY/Klinefelter syndrome. Am J Med Genet C Semin Med Genet. 2020 Jun;184(2):327-333. doi: 10.1002/ajmg.c.31784. Epub 2020 Jun 16. PMID 32542985
- See also: KS&A supports individuals with XXY/Klinefelter syndrome and other X&Y chromosome variations — http://www.genetic.org
- See also: The eXtraordinary Kids Clinic at Children's Hospital Colorado is a multispecialty clinic that evaluates and treats children, adolescents, and young adults with all X&Y chromosome variations — http://www.childrenscolorado.org/conditions/behavior/xychromosome.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone Gel 1% | Placebo Gel
Started | 28 | 20
Completed | 26 | 18
Not Completed | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Gel 1% | Placebo Gel | Total
Number analyzed (Participants) | 28 | 20 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 20 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.23 (1.15) | 12.22 (1.55) | 12.22 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 20 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 25 | 19 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 17 | 40
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 18 | 46
  Canada | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Delis-Kaplan Executive Function System
Description: A collection of subtests from the Delis-Kaplan Executive Function System will be used to evaluate different domains of executive functions including planning, problem solving, fluency, inhibition, and working memory. Possible scaled scores range from 0-20 (mean of 10), with higher scores indicating better performance. The value of the change in scaled score from baseline is reported.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: Variability in participants analyzed for each outcome measure is due to participant inability to complete the measure or missing study visits.
Measure: Mean (Standard Deviation); unit: Scaled scores
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 25 | 17
Scaled scores
  Verbal Fluency | -0.72 (2.35) | 1.29 (3.0)
  Color-Word Interference | 1.28 (3.1) | 0.65 (2.71)
  Sorting | 0.75 (3.24) | 0.76 (1.82)
  20 Questions | 0.60 (2.99) | 1.59 (4.06)

2. Primary Outcome: Change From Baseline on the Bruininks-Oseretsky Test of Motor Development - 2
Description: This test evaluates many aspects of motor functioning including fine and gross motor skills, visual motor integration, motor planning, and motor coordination. Possible scores range from 20-80, with higher scores indicating a better outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 26 | 17
score on a scale
  Baseline | 39.92 (7.55) | 35.52 (6.38)
  1 Year | 41.34 (7.96) | 37.17 (6.6)

3. Primary Outcome: Change From Baseline on the Conners Parent Rating Scales: DSM Attention
Description: This questionnaire allows parents to rate many aspects of behavior including attention, hyperactivity, anxiety, social skills, and emotional lability. The range of possible scores is 0 to 100 (Mean T-score 50), with higher scores indicating a worse outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 26 | 18
score on a scale
  Baseline | 64.2 (10.6) | 62.8 (8.8)
  1 Year | 58.1 (11.4) | 59.3 (12.1)

4. Primary Outcome: Change From Baseline on the Conners Parent Rating Scales: DSM Hyperactivity
Description: as for outcome 3
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 26 | 18
score on a scale
  Baseline | 60.7 (10.7) | 57.2 (10.1)
  1 Year | 53.4 (10.5) | 54.4 (11.5)

5. Primary Outcome: Change From Baseline on the Conners Parent Rating Scales: Anxiety
Description: as for outcome 3
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 25 | 17
score on a scale
  Baseline | 59.7 (12.7) | 62.2 (13.7)
  1 Year | 54.0 (10.4) | 62.8 (18.8)

6. Primary Outcome: Change From Baseline on the Conners Parent Rating Scales: Social Skills
Description: This questionnaire allows parents to rate many aspects of behavior including attention, hyperactivity, anxiety, social skills, and emotional lability. The range of possible scores is 0 to 100, with higher scores indicating a worse outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 26 | 17
score on a scale
  Baseline | 64.3 (14.0) | 66.4 (14.6)
  1 Year | 62.7 (14.6) | 63.2 (15.0)

7. Primary Outcome: Change From Baseline on the Conners Parent Rating Scales: Emotional Lability
Description: as for outcome 6
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 25 | 17
score on a scale
  Baseline | 59.4 (14.1) | 61.3 (16.4)
  1 Year | 57.3 (13.9) | 54.4 (18.1)

8. Secondary Outcome: Change From Baseline on the Vineland Adaptive Behavior Scales - 2nd Edition
Description: The Vineland-2 is an interview evaluating adaptive skills in the areas of communication, daily living skills, social skills, and motor skills. Possible scores range from 20 to 160 (mean 100), with higher scores indicating a better outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 25 | 14
score on a scale
  Baseline | 78.7 (8.6) | 75.8 (10.3)
  Change at 1 year | 82.2 (9.8) | 78.4 (11.2)

9. Secondary Outcome: Change From Baseline on the Wechsler Intelligence Scale for Children - Fourth Edition
Description: This standardized assessment of cognitive functioning allows for evaluation of verbal and nonverbal cognitive skills, working memory, and processing speed. Possible full scale IQ scores range from 40-180 (mean 100), with higher scores indicating a better outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 24 | 17
score on a scale
  Baseline | 86.8 (16.1) | 83.9 (14.1)
  1 Year | 88.7 (18.8) | 84.6 (15.1)

10. Secondary Outcome: Change From Baseline on the Comprehensive Test of Phonological Processing
Description: This standardized test evaluates reading and language skills. Possible scores range from 20-200 (Mean Standard Score 100), with higher scores indicating a better outcome.
Time Frame: Visit 1 (baseline) and Visit 5 (1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Gel 1% | Placebo Gel
Number analyzed (Participants) | 24 | 16
score on a scale
  Baseline | 77.0 (14.1) | 78.1 (15.9)
  Change at 1 Year | 77.1 (14.3) | 77.4 (17.8)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Testosterone Gel 1% | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/20
Other Adverse Events (participants affected / at risk) | 25/28 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel 1% (N=28) | Placebo Gel (N=20)
Acne (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Behavioral agitation (Psychiatric disorders) | 10 (10) | 5 (5)
Skin reaction at application site (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Gynecomstia (Endocrine disorders) | 1 (1) | 2 (2)
Scrotal Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Low White Blood Cell count (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Advance bone age >1 year (Musculoskeletal and connective tissue disorders) | 13 (13) | 4 (4)
Transaminase elevation >ULN (Hepatobiliary disorders) | 25 (25) | 15 (15)
Testosterone effects in female caregiver (Endocrine disorders) | 2 (2) | 1 (1)
Elevated Triglycerides >250mg/dL (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
BASC-2 Critical Item change (Psychiatric disorders) | 13 (13) | 9 (9) — BASC-2 Critical items related to psychiatric symptoms (depression, self-esteem) newly endorsed or increased from baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT01585831/Prot_SAP_000.pdf